CLINICAL TRIAL: NCT04105101
Title: The Effect of a Novel Passive Shoulder Exoskeleton on the Human Body During Simulated Industrial Tasks
Brief Title: The Effect of a Novel Passive Shoulder Exoskeleton During Industrial Work
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Principal investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EXOTEST2019
Record Dates: First submitted 2019-09-19; First posted 2019-09-26 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Exoskeleton Device
Keywords: Human-centered robotics; Prototype evaluation; Industry

STUDY DESIGN:
Intervention Model Description: Randomized counterbalanced cross-over design
Who Masked: Participant
Masking Description: Blinding is not possible in this testing set-up, participants however are not informed about the exact purpose of the tests and which exoskeleton is a prototype and which exoskeleton is a commercially available exoskeleton.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prototype exoskeleon (Experimental): The experimental trial will be performed with the prototype exoskeleton
  Interventions: Device: Industrial passive shoulder exoskeleton
- Skel-Ex (Experimental): The experimental protocol will be performed with the commercially available Skel-Ex 360 (Skel-Ex, Rotterdam, The Netherlands)
  Interventions: Device: Industrial passive shoulder exoskeleton
- No exoskeleton (Experimental): The experimental protocol will be performed without exoskeleton.
  Interventions: Device: Industrial passive shoulder exoskeleton

INTERVENTIONS:
Device: Industrial passive shoulder exoskeleton — Both exoskeleton types are passive shoulder exoskeletons. The goal is to compare the human response to the simulated industrial tasks between the different exoskeleton conditions.

SUMMARY:
After designing a first prototype of next generation industrial exoskeleton, the system should be evaluated in laboratory conditions. In order to evaluate the passive shoulder exoskeleton, designed to assist workers, a protocol is developed in which parts of industrial work is simulated. The results of this evaluation will serve as input for the next iterative design process/cycle of the prototype.

In this study 15 subjects will be recruited. During a 3.5h lab visit, each subject will perform three identical experimental trials; one trial without exoskeleton, one trial with a commercially available exoskeleton and one with the newly developed prototype. To avoid sequence bias, the order of the trials will be randomized (counterbalanced). The protocol consists of 6 tasks, always performed in the same sequence; lifting 5 kg 5 times from hip height to overhead height, completing a wiring task overhead (90 sec), 6 minutes walking, 6 min lifting from hip to overhead height (10 kg), 6 min lifting from ground to hip level (10 kg) and drilling for 30 sec with a force of 60N (±20 N). Before each task, 5 min of rest will be provided, and the subject will receive 10 min of rest in between different experimental trials. Electrocardiographic data, chest expansion and skin temperature will be monitored through a belt (Equivital, AD Instruments). An ergospirometric device (K5, Cosmed) will be used to gather gas exchange data, and (non-invasive) EMG electrodes will be applied to collect muscle activity data during the trials (Cometa). IMUs will be applied to the subjects' extremities to analyse the movement pattern (Technaid). Furthermore, questionnaires will be filled out to assess the subjective experience (Rating of Perceived Exertion, Sustained Usability Scale, Local Discomfort Scale).

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals (based on ParQ questionnaire)

Exclusion Criteria:

* work related disorders
* shoulder injuries in the past
* back injuries in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Surface electromyography | Electromyographic data will be collected continuously during all simulated industrial tasks. This will take 3 hours in total.
  Cometa (mini wave) sensors with Ambu (BlueSensor) electrodes will be used to collect electromyographic data conform the SENIAM guidelines. The muscles that will be monitored are: erector spinae, biceps femoris, rectus femoris, gastrocnemius, tibialis anterior, trapezius (all three parts), deltoideus (all three parts), pectoralis major, latissimus dorsi, brachioradialis, biceps brachii, triceps brachii on both the left and the right side of the body. The locations of the sensors will be prepared by shaving, abrasion with sandpaper and cleaning with alcohol. To allow relative expression of muscle activities, maximal voluntary isometric contractions (MVIC) of each muscle that is being monitored will be collected. The average of the maximal activity out of the best two out of three contractions will serve as the MVIC value. The outcomes will be the activities of the muscles (as a percentage of the MVIC) monitored during the tests.
Heart rate | Heart rate will be monitored continuously during all tasks. This will take 3 hours in total
  An Equivital belt will be worn by all subject. heart rate can be computed from the ECG signal
Metabolic cost | Metabolic cost will be monitored continuously during all tasks. This will take 3 hours in total
  A Cosmed K5 device will be used to measure oxygen consumption and carbon dioxide exhaust during every task lasting longer than three minutes. The outcome measures are the metabolic cost during walking, overhead lifting and lower lifting. The metabolic cost will be computed with the measured oxygen consumption and carbon dioxide exhaust.
session Rating of Perceived exertion | the sRPE will be asked at the end of the task. The entire protocol will last for approximately 3 hours.
  This questionnaire scores the perceived exertion during a task. Scores can range from 6 to 20, with 6 being not exhausted at all and 20 being extremely exhausted. The scale is only one question, so no sub-scales are available

SECONDARY OUTCOMES:
Heart rate variability | Will be computed for every task. The recording will be continuous throughout the whole protocol, lasting for approximately 3 hours.
  The distance between R peaks in the electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Romain Meeusen, Prof. dr., Principal Investigator — VUB
Locations (1):
- Lichamelijk Opvoeding en Kinesitherapie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
The data can not be made public as this is part of a larger project